CLINICAL TRIAL: NCT00974389
Title: Phase II Study of Combination Chemotherapy With S-1 Plus Avastin in Unresectable or Recurrent Colorectal Cancer After Failure of Prior Chemotherapy, Including Irinotecan and Oxaliplatin Regimens.
Brief Title: S-1 and Bevacizumab in Treating Patients With Colorectal Cancer That is Recurrent or Cannot Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka Medical College (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: OSAKA-TRICC0901; CDR0000649021 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-09

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage III rectal cancer; stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Biological: bevacizumab
Drug: tegafur-gimeracil-oteracil potassium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as S-1, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving S-1 together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving S-1 together with bevacizumab works as third-line therapy in treating patients with colorectal cancer that is recurrent or that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate giving S-1 with bevacizumab to see how well it works as third-line therapy in KRAS-mutation patients with unresectable or recurrent colorectal cancer.

OUTLINE: Patients receive oral S-1 twice daily on days 1-28 and bevacizumab IV on days 1, 15, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal carcinoma

  * Inoperable, locally advanced, or metastatic disease
  * KRAS-mutated
* Concurrently receiving treatment containing irinotecan and oxaliplatin regimens for unresectable or recurrent colorectal cancer
* Measurable disease according to RECIST
* No moderate or severe ascites or pleural effusion requiring treatment
* No metastasis to the CNS

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* White blood cell count > 3,500/mm³ but < 12,000/mm³
* Neutrophil count > 1,500/mm³
* Hemoglobin > 9.0 g/dL
* Platelet count > 100,000/mm³
* Total bilirubin < 1.5 mg/dL
* AST and ALT < 100 U/L (< 200 U/L in patients with liver metastasis)
* Serum creatinine < 1.2 mg/dL
* Creatinine clearance ≥ 50 mL/min
* Urine dipstick for proteinuria < 1+
* INR < 1.5
* Not pregnant or nursing
* Able to take capsules orally
* No active second cancer
* No active infections (e.g., patients with pyrexia of ≥ 38°C)
* No serious complications (e.g., pulmonary fibrosis, interstitial pneumonitis, heart failure, renal failure, hepatic failure, poorly controlled diabetes, or hypertension)
* No electrocardiographic abnormalities with cardiac disorder that would clinically preclude the execution of the study as judged by the investigator
* No serious drug hypersensitivity or a history of drug allergy
* No thrombosis, cerebral infarction, myocardial infarction, or pulmonary embolism
* No history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* No clinically significant traumatic injury within the past 4 weeks
* No severe mental disorder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent low-dose aspirin therapy (< 325 mg/day) allowed
* More than 4 weeks since prior major surgical procedure or open biopsy
* No prior therapy radiotherapy
* No prior therapy with S-1
* No prior chemotherapy include irinotecan and oxaliplatin as first- or second-line treatment.
* No concurrent continuous treatment with steroids
* No concurrent treatment with flucytosine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Disease-control rate

SECONDARY OUTCOMES:
Response rate
Progression-free survival
Overall survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Hiroya Takiuchi, MD, PhD, Principal Investigator — Osaka Medical College
Locations (1):
- Osaka Medical College, Takatsuki, Osaka, Japan